CLINICAL TRIAL: NCT06876883
Title: MItral Regurgitation Risk Assessment and CLinical modElling (MIRACLE Study)
Brief Title: MItral Regurgitation Risk Assessment and CLinical modElling
Acronym: MIRACLE
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Principle Investigator, Sun Yat-sen University
Other Study IDs: MIRACLE study
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Mitral Insufficiency; Mitral Regurgitation (MR)
Keywords: mitral regurgitation; all-cause mortality; clinical modelling; cardiovascular mortality; heart failure hospitalization
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MR: Patients with ≥ moderate mitral regurgitation

SUMMARY:
Mitral regurgitation (MR) is a common valvular heart disease worldwide, and untreated severe MR is associated with an elevated risk of heart failure and mortality. According to causes, MR could be divided into primary or secondary MR. The risk factors of mortality or heart failure hospitalization in different types of MR patients are under intensive investigation.

MItral Regurgitation risk Assessment and CLinical modElling (MIRACLE) study is a prospective cohort study including adult patients diagnosed with ≥ moderate MR during hospitalization. Comprehensive echocardiographic examination was conducted at baseline evaluating valvular heart disease severity, atrial and ventricular systolic/diastolic function, pulmonary artery systolic pressure (PASP), etc. We aim to evaluate the prognostic risk factors of patients with MR and construct a prognostic clinical model to guide clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ≥ moderate mitral regurgitation during hospitalization.
* Aged over 18 yrs.

Exclusion Criteria:

* Patients unable to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with ≥ moderate mitral regurgitation (MR) during hospitalization were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-06-15 (Actual); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, an average of 5 years
  Death due to any cause after enrollment

SECONDARY OUTCOMES:
Cardiovascular mortality | Through study completion, an average of 5 years
  Death due to cardiovascular causes, including heart failure, myocardial infarction, fatal arrhythmia, major bleeding, stroke, sudden death and thromboembolism.
Heart Failure Hospitalization (HFH) | Through study completion, an average of 5 years
  Hospitalization with the primary reason for admission as acute decompensated HF and administration of intravenous or mechanical heart failure therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen Univerity, Guangzhou, Guangdong, China